CLINICAL TRIAL: NCT06714942
Title: Efficacy and Safety of a Proprietary Blend of Ashwagandha Root Extract (Aqueous) in Adult Men and Women With High Stress and Anxiety: A Randomized, Double-blind, Three-arm, Parallel, Placebo-controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Agaja Pharma Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGJ-1051-2023-01
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): One capsule of Proprietary Blend of Ashwagandha 300 mg twice a day, orally with water.
  Interventions: Dietary Supplement: Proprietary Blend of Ashwagandha
- Comparator Group (Experimental): One capsule of KSM-66 Ashwagandha 300mg two times a day, orally with water
  Interventions: Dietary Supplement: KSM-66 Ashwagandha root extract
- Control Group (Placebo Comparator): One capsule of Placebo two times a day, orally with water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Proprietary Blend of Ashwagandha — One capsule (300mg) is taken twice daily with water
  Arms: Treatment Group
Dietary Supplement: KSM-66 Ashwagandha root extract — One capsule (300mg) is taken twice daily with water
  Arms: Comparator Group
Dietary Supplement: Placebo — One capsule (300mg) is taken twice daily with water
  Arms: Control Group

SUMMARY:
This is a Multi-center, Multi-national, Prospective, Randomized, Double-Blind, Placebo- Controlled three arm study to evaluate the efficacy and safety of a Proprietary Blend of Ashwagandha Root Extract (Aqueous) in Adult Men and Women with High Stress and Anxiety. All eligible subjects who meet the Inclusion and Exclusion criteria will be part of the study. Subjects will be informed about the purpose of the study and signed informed consent will be taken. Subjects will be randomized to either one of the three treatment arms. Subjects will then be asked to either take one capsule containing the proprietary blend of Ashwagandha root extract or Ashwagandha root extract or Placebo orally twice daily with a glass of water for 8 weeks. The primary objective is to compare the efficacy of a proprietary blend of Ashwagandha root extract in adults experiencing stress and anxiety. The secondary objective is to compare the safety of a proprietary blend versus KSM-66 versus Placebo in adults experiencing stress and anxiety.

DETAILED DESCRIPTION:
To qualify for the study, participants must be aged between 18 to 55 years experiencing signs and symptoms suggestive of stress (e.g., difficulty, concentrating, physical exhaustion, anxiety, restlessness, insomnia, headache, fatigue, loss of appetite, worry, sweating, mental confusion, etc.).

In this study, a maximum of 51 patients will be enrolled and the goal is to complete the study with at least 45 patients.

After signing this consent form, participants will answer questions regarding their medical history, including any medications they are taking. Physical exams with vital signs (pulse, temperature, sitting blood pressure and respiratory rate) will be performed at both visits by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist, or Medical Doctor.

A blood sample will be required from subjects. Subject's right or left arm will be used as the blood draw site, requiring a 5mL sample.e blood will be analyzing Cortisol level. These blood draws will be administered by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist or Medical Doctor.

A two-page Hamilton Anxiety Rating Scale (HAM-A) Test and Perceived Stress Scale (PSS) will be given and administered as self-assessment.

All eligible participants, will be given the required quantity of the study medication for self-administration, sufficient till the Visit 3- End of study visit, 8 weeks ± 4 Days. Participants will be randomized to either one of the three treatment arms.

Participants will be instructed to take one capsule of study medication to which they are randomized twice daily, with ambient temperature water for 8 weeks at home. Participants will be asked to visit the site for Visit 2 (4 weeks ± 4 Days), Visit 3 (8 weeks ± 4 Days). Adverse events and concomitant medication will be recorded throughout the study. Participants will be asked to get used and unused study medications and their subject diaries in this visit. All the participants will be asked to continue their routine diet and physical activities during the whole study period.

The primary end point is mean change in serum cortisol level from baseline. The secondary end points are Perceived Stress Scale (PSS) questionnaire, Hamilton Anxiety Rating Scale (HAM-A) questionnaire, Profile of Mood States (POMS, abbreviated version) questionnaire, Oxford Happiness Questionnaire from baseline. The safety end points are the Number and proportion of Treatment-Emergent Adverse Events (TEAEs) over 8 weeks and the Number and proportion of Treatment-Emergent Serious Adverse Events (TESAE) over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (male and female) aged between 18 and 65 years.
2. Experiencing signs and symptoms suggestive of stress (e.g., difficulty, concentrating, physical exhaustion, anxiety, restlessness, insomnia, headache, fatigue, loss of appetite, worry, sweating, mental confusion, etc.).
3. Hamilton Anxiety Rating Scale (HAM-A) total score between 14 and 30 at the screening/randomization visit.
4. Perceived Stress Scale (PSS) score ≥13 at the screening/randomization visit.
5. BMI between 20 and 35.
6. No plan to commence new treatments over the study period.
7. Medication-free (any medications are known to affect stress and anxiety) for at least 4 weeks. Use of analgesics (once a week) or contraceptive pills are permissible.
8. Must have the ability and willingness to sign an informed consent and to comply with all study procedures.

Exclusion Criteria:

1. Patients receiving any of the medications known to affect stress and anxiety (corticosteroids, antidepressants, antipsychotics, mood stabilizers, and anti-epileptic medications) during 4 weeks prior to screening.
2. Patients having a total score of less than 14 on HAM-A at screening.
3. Patients currently (or within the past 4 weeks prior to screening) taking any over-the-counter use of herbal extracts such as Ginkgo Biloba, St. John's Wort, Omega-3, etc.
4. Patients with a depressive episode, suicidal tendency, panic disorder, social phobia, obsessive-compulsory disorder; alcohol dependency; schizophrenia, and mania.
5. Patients with known post-traumatic stress disorder (PTSD) and Generalized Anxiety Disorder (GAD).
6. Patients who have an established practice of meditation and relaxation techniques for three or more months.
7. Patients with known clinically significant acute unstable hepatic, renal, cardiovascular, or respiratory disease that will prevent participation in the study.
8. Patients with a history of alcohol, tobacco dependence, or any substance abuse.
9. Pregnant and lactating women or suspected to be pregnant.
10. Patients with known hypersensitivity to Ashwagandha.
11. Patients who had participated in other clinical trials during the previous 3 months.
12. Patients who have any clinical condition, according to the investigator who does not allow safe fulfilment of clinical trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
Serum cortisol level | Blood samples for serum cortisol will be collected at Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1) and Visit 3- (Week 8)]

SECONDARY OUTCOMES:
Perceived Stress Scale Score (PSS) | PSS assessment will be done at Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4), and Visit 3 (Week 8).
  The Perceived Stress Scale (PSS-10) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. The questions in the PSS ask about feelings and thoughts during the last month.
Hamilton Anxiety Rating Scale (HAM-A) | HAM-A assessment will be done at Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4), and Visit 3 (Week 8).
  The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms and is still widely used today in both clinical and research settings. The HAM-A scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Profile of Mood States (POMS, abbreviated version) | POMS assessment will be done at Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4), and Visit 3 (Week 8).
  The POMS is a 40-item questionnaire rated on a 5-point Likert Scale, asking respondents how they feel right now. Scores are calculated for Tension, Anger, Fatigue, Depression, Esteem-related affect, Vigor, Confusion, and Total Mood Disturbance.
Oxford Happiness Questionnaire | Oxford Happiness Questionnaire assessment will be done at Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4), and Visit 3 (Week 8).
  The Oxford Happiness Scale (OHS) is a psychological assessment tool designed to measure an individual's subjective level of happiness. It was developed by researchers Michael Argyle and Peter Hills at the University of Oxford. The scale is widely used in positive psychology and well-being research to evaluate happiness as a multidimensional concept, encompassing emotional, cognitive, and social aspects.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided